CLINICAL TRIAL: NCT04758195
Title: A Prospective, Randomized, Open, Parallel Trial of Transanal Irrigation to Prevent Major Low Anterior Resection Syndrome in Rectal Cancer Patients
Brief Title: Transanal Irrigation to Prevent Major Low Anterior Resection Syndrome
Acronym: TAILARS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: E2021004
Record Dates: First submitted 2021-02-15; First posted 2021-02-17 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Low Anterior Resection Syndrome
Keywords: Low Anterior Resection Syndrome; Transanal irrigation; Rectal cancer; Prevention
MeSH Terms: conditions — Low Anterior Resection Syndrome; Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transanal irrigation (Experimental): Transanal irrigation (TAI) is performed using the irrigation bag, electronic irrigation system, or balloon catheter with syringe. TAI is performed with up to 2000 ml tap water every 24-48 hours (3-7 times per week) over the course of 6 months.
  Interventions: Procedure: Transanal irrigation
- Best supportive therapy (Active Comparator): Best supportive therapy consists of dietary modification, pelvic floor muscle training, biofeedback, and necessary medication.
  Interventions: Other: Best supportive therapy

INTERVENTIONS:
Procedure: Transanal irrigation — Transanal irrigation (TAI) is performed using the irrigation bag, electronic irrigation system, or balloon catheter with syringe. TAI is performed with up to 2000 ml tap water every 24-48 hours (3-7 times per week) over the course of 6 months.
  Arms: Transanal irrigation
Other: Best supportive therapy — Best supportive therapy consists of dietary modification, pelvic floor muscle training, biofeedback, and necessary medication.
  Arms: Best supportive therapy

SUMMARY:
Bowel dysfunction after rectal cancer resection comprises a vast array of bowel symptoms and associated quality-of-life impairment, collectively termed as low anterior resection syndrome (LARS). There are 40%-60% patients who suffer from major LARS after sphincter-preserving surgery. No consensus exists for LARS treatment or prevention. Transanal irrigation (TAI) was reported to play a helpful role in the management of major LARS and fecal incontinence. However, the preventive effect and daily accessibility need further confirmation. In this randomized trial, TAI compared with best support treatment, is used in patients who received curative low anterior resection for rectal cancer with diverting stoma, after completion of the stoma reversal. The primary outcome is the occurrence of major LARS after 6 months of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-75 years old
* Curative low anterior resection for rectal cancer with diverting stoma
* Stoma closure within 1 month
* Preoperative radiotherapy or height of anastomosis less than 5 cm from anal verge
* No evidence of anastomotic leakage or severe stenosis

Exclusion Criteria:

* Tumor recurrence or distant metastasis
* Secondary operation with stoma
* Prior disease impairing bowel function except for rectal cancer
* Any contraindication for transanal irrigation
* Pregnant or nursing
* Serious cardiovascular disease, uncontrolled infections, or other serious uncontrolled concomitant disease
* Cognitive or psychological disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with major low anterior resection syndrome score (LARS score) | at the time of 6 months since the start of treatment

SECONDARY OUTCOMES:
Quality of life impairment assessed by Short Form 36 (SF-36) | at the time of 6, 12 months since the start of treatment
  Quality of life will be assessed by Short Form 36 (SF-36) health questionnaire.
Number of participants with major low anterior resection syndrome score (LARS score) | at the time of 1, 3, 12 months since the start of treatment
Bowel function impairment | at the time of 6, 12 months since the start of treatment
  Bowel function will be assessed by Memorial Sloan Kettering Cancer Centre Bowel Function Instrument (MSKCC BFI). Stool frequency will be recorded in the day and night.
Fecal continence impairment | at the time of 6, 12 months since the start of treatment
  Fecal incontinence will be assessed by Wexner incontinence scale.

OTHER OUTCOMES:
Anorectal function impairment | at the time of 6 months since the start of treatment
  Anorectal function will be assessed by anorectal manometry.

CONTACTS AND LOCATIONS:
Overall Officials: Qiyuan Qin, M.D., Principal Investigator — The Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China